CLINICAL TRIAL: NCT06834607
Title: Physician Modified Endovascular Grafts for the Treatment of Elective, Symptomatic or Ruptured Complex Aortic Aneurysms
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Akhilesh Jain (Other)
Responsible Party: Sponsor-Investigator, Akhilesh Jain, Chief of Vascular Surgery, Harford Hospital, Hartford Hospital
Organization: Hartford Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ref #: 040115; G250012 (Other: U.S. Food & Drug Administration)
Record Dates: First submitted 2025-02-10; First posted 2025-02-19 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Juxta Renal Abdominal Aortic Aneurysm Without Rupture; Complex Aortic Aneurysms; Aortic Aneurysm
Keywords: Physician Modified Endograft; PMEG; Complex aortic aneurysms; Juxta renal aortic aneurysm
MeSH Terms: conditions — Aortic Aneurysm

STUDY DESIGN:
Intervention Model Description: Prospective, single center, nonrandomized, single arm study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Treatment arm (Experimental)
  Interventions: Device: Physician Modified Aortic Endograft repair for complex aortic aneurysm

INTERVENTIONS:
Device: Physician Modified Aortic Endograft repair for complex aortic aneurysm — To assess the use of the Physician-Modified Endovascular Grafts to repair juxtarenal aneurysms in high-risk subjects considered to be unsuitable candidates for open surgical repair, have limited or no other options for treatment, and having appropriate anatomy.

SUMMARY:
The primary objective of the clinical investigation "Physician Modified Endovascular Grafts for the Treatment of Elective, Symptomatic or Ruptured Complex Aortic Aneurysms" is to assess the use of the Physician-Modified Endovascular Grafts to repair juxtarenal aneurysms in high-risk subjects considered to be high risk candidates for open surgical repair, have limited or no other options for on label treatment with an FDA approved device, and having appropriate anatomy.

DETAILED DESCRIPTION:
The primary intent of the study is to assess safety and preliminary effectiveness of the physician modified endografts acutely (i.e., treatment success and technical success), at 30 days (i.e., the rate of major adverse events (MAE)) and at 6 months, 12 months and annually to 5 years (i.e., the proportion of treatment group subjects that achieve and maintain treatment success).

ELIGIBILITY:
Inclusion Criteria:

1. Patient is ≥ 18 years of age
2. Patients who are male or non-pregnant female (females of child bearing potential must have a negative pregnancy test prior to enrollment into the study)
3. Patient or Legally Authorized Representative has signed an Institutional Review Board (IRB) approved Informed Consent Form
4. Patient has a juxtarenal abdominal aortic aneurysm that meets at least one of the following:

   1. An aneurysm with a maximum diameter of ≥ 5.5 cm for male (≥ 5.0 cm for female) or 2 times the normal diameter just proximal to the aneurysm using orthogonal (i.e., perpendicular to the centerline) measurements
   2. Aneurysm with a history of growth > 0.5 cm in 6 months
   3. Saccular aneurysm deemed at significant risk for rupture
   4. Symptomatic aneurysm
   5. Ruptured aneurysm
5. Patient has patent iliac or femoral arteries, with or without the use of conduit, that will allow endovascular access with the physician modified endovascular graft.
6. Patient has a suitable non-aneurysmal proximal aortic neck of ≥ 2 mm inferior to the most distal renal artery ostium.
7. Patient has a suitable non-aneurysmal distal iliac artery length (seal zone) of ≥ 15mm. The resultant repair should preserve patency in at least one hypogastric artery.
8. Patient has a suitable non-aneurysmal proximal aortic neck diameter between 20 and 32 mm, averaged across the diameters at the Celiac, SMA, at the lowest patent renal artery and at the midpoint of the renal arteries.
9. Patient has suitable non-aneurysmal distal common iliac diameters between 8 and 20 mm.
10. Patient has juxtarenal aortic neck angulation ≤ 60°
11. Target branch vessel diameter ≥ 5 mm.
12. Patient must be willing to comply with all required follow-up exams.

Exclusion Criteria:

1. Patient has a mycotic aneurysm or has an active systemic or local infection that may increase the risk of endovascular infection
2. Patient has unstable angina (defined as angina with a progressive increase in symptoms, new onset at rest or nocturnal angina, or onset of prolonged angina)
3. Patient has a major surgical or interventional procedure, not related to the endovascular repair, planned within +/- 30 days of the AAA repair.
4. Patient has history of an aortopathic connective tissue disease (e.g. Marfan's or Ehler's-Danlos syndrome).
5. Patient has a known hypersensitivity or contraindication to anticoagulation or contrast media that is not amenable to pre-treatment.
6. Patient has known allergy or intolerance to stainless steel, nitiol, or gold (gold-plated tungsten)
7. Patient has a body habitus that would inhibit X-ray visualization of the aorta
8. Patient has a limited life expectancy of less than 1 year
9. Patient is currently participating in another investigational device or drug clinical trial
10. Patient has other medical, social or psychological conditions that, in the opinion of the investigator, preclude them from receiving the pre-treatment, required treatment, and post-treatment procedures and evaluations.
11. Thrombus or excessive calcification within the neck of the aneurysm
12. Branch vessel stenosis ≥ 80 %
13. Patients treatable on label with FDA approved EVAR or FEVAR device and can wait for device availability.
14. Subject is willing and eligible to enroll in a manufacturer-sponsored study at the investigational site, or the subject is willing and eligible to participate in a study with a manufacturer-made device at another institution.

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2032-05-01 (Estimated)

PRIMARY OUTCOMES:
Primary Safety Endpoint: Safety of PMEG device will be measured by proportion of subjects who experience a Major Adverse Event (MAE) within 30 days of the index procedure. | 30 days
  The Primary Safety Endpoint is defined as the proportion of subjects who experience a Major Adverse Event (MAE) within 30 days of the index procedure.
  Major Adverse Events that will be recorded include the following:
  * All-cause mortality
  * Myocardial Infarction
  * Stroke
  * Renal Failure
  * Respiratory Failure
  * Paraplegia
  * Bowel Ischemia
  * Procedural Blood Loss (> 1000cc)
Primary Effectiveness Endpoint: Will be measured by calculating the proportion of patients that achieve Treatment Success | 12 months
  Effectiveness of the PMEG device will be measured by the calculating the proportion of subjects that achieve Treatment Success.
  Treatment Success is a will be assessed at 12 months and is define by a combination of following criteria to be met:
  * Technical Success (at the index procedure).
  * Freedom from Type I & III endoleaks at 12 months
  * Freedom from stent graft migration at 12 months
  * Freedom from aortic aneurysm enlargement at 12 months
  * Freedom from aortic aneurysm rupture and conversion to open repair through 12 months
  Technical Success at the index procedure will be defined by: The physician was able to insert the delivery catheter and deliver the physician modified endovascular graft to the treatment site and preserve blood flow into the vessels intended to have blood flow preserved.

SECONDARY OUTCOMES:
Secondary Safety Endpoints: Will be assessed by measuring proportion of patients encountering any of the following adverse events | Through 5 years
  The adverse events will be evaluated at 30 days, 6 months, 12 months following the initial implant procedure and annually through 5 years.
  The adverse events to be evaluated include:
  * Mortality
  * Aneurysm related mortality
  * Aneurysm rupture
  * Major Adverse Events (MAE)
  * Renal Failure with or without permanent dialysis
  * Graft infection
Secondary Effectiveness Endpoints: Defined by proportion of patients experiencing the following events. | Through 5 years
  The secondary effectiveness endpoints will be evaluated at 30 days, 6 months, 12 months following the initial implant procedure and annually through 5 years:
  Following secondary endpoints will be evaluated for every patient:
  * Technical Success (evaluated at 30-days)
  * Stent graft migration (>10 mm)
  * All endoleaks, including Type I & III endoleaks
  * AAA enlargement
  * Patency related events
  * Device integrity failure
  * Conversion to open repair
  * Secondary intervention (reason and type)

CONTACTS AND LOCATIONS:
Locations (1):
- Hartford Hospital, Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No